CLINICAL TRIAL: NCT03469401
Title: Evaluation of the Detection of B D Glucan in Peritonitis Fluid in Intensive Care Unit (ICU) Patients With Peritonitis for the Diagnosis of Fungal Peritonitis, Compared to Routine Microbiology Diagnosis Method. The PERICAND Study
Brief Title: Evaluation of BD Glucan in Peritoneal Fluid for the Diagnosis of Fungal Peritonitis
Acronym: PERICAND
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0775
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Adult Patient (Over 18 Yr-old) Admitted to the ICU for Acute Peritonitis
MeSH Terms: interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peritoneal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- intervention: Adult patient (over 18 yr-old) admitted to the ICU for acute peritonitis with a peritoneal fl:uid sample obtained via surgery or radiological drainage
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Evaluation of sensibility, specificity, negative and positive predictive value of BD glucan in peritoneal fluid for diagnosis of fungal peritonitis, compared with fungal culture

SUMMARY:
Invasive candidiasis has a high mortality rate, around 40%. Outcome remains tightly linked to the time of treatment administration. Routine microbiological techniques give results too lately to allow prompt antifungal therapy initiation (at least 48 hours). It is important to develop diagnostic tools to initiate antifungal therapy as early as possible.

The B D glucan detection, one of the major components of the candida cell wall, can be useful for a early diagnosis.

There are several techniques on the market for the detection of glucan. In Europe and America, the most used is Fungitell (Associated of Cape Cod, Inc).

There is several studies about the use of such kits for fungemia. A number of studies are reporting evidences of a early diagnosis.

But, in medical literature, there isn't study focused on the detection of B D glucan in peritoneal fluid for Candida peritonitis diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* written informed consent for inclusion in the study
* stay in intensive care unit
* diagnosed with a peritonitis
* peritoneal fluid collected by a surgery or radiology procedure, analysed at bacteriology laboratory of l'institut des agents infectieux, l'hôpital de la Croix Rousse

Exclusion Criteria:

* Pregnant woman
* Moribund patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (over 18 yr-old) admitted to the ICU for acute peritonitis
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of sensibility, specificity, negative and positive predictive value of BD glucan in peritoneal fluid for diagnosis of fungal peritonitis, compared with fungal culture | 1 year
  Evaluation of sensibility, specificity, negative and positive predictive value of BD glucan in peritoneal fluid for diagnosis of fungal peritonitis, compared with fungal culture

CONTACTS AND LOCATIONS:
Overall Officials: Florent WALLET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nourry E, Wallet F, Darien M, Menotti J, Dupont D, Allaouchiche B, Argaud L, Richard JC, Guichon C, Rimmele T, Bohe J, Thiollere F, Vassal O, Lepape A, Wallon M, Persat F, Friggeri A. Use of 1,3-Beta-D-Glucan concentration in peritoneal fluid for the diagnosis of intra-abdominal Candidiasis in Critically-ill patients. Med Mycol. 2023 Mar 20:myad029. doi: 10.1093/mmy/myad029. Online ahead of print. PMID 36941133